CLINICAL TRIAL: NCT06055335
Title: EVALUATION OF LUNG DYNAMICS AND RESPIRATORY FUNCTIONS IN PATIENTS APPLIED WITH MINIMAL FLOW ANESTHESIA: A PROSPECTIVE, RANDOMIZED STUDY
Brief Title: Assessing Lung Dynamics and Respiratory Functions in Minimal Flow Anesthesia: A Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Erkan Cem ÇELİK, Associate Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2/106 25.03.2021
Record Dates: First submitted 2023-09-14; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Medium Flow Anesthesia; Minimal Flow Anesthesia; Pulmonary Function Test; Compliance, Patient; Peak Inspiratuar Pressure
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medium flow anesthesia (Experimental): After reaching the MAC 1 value with 4lt/min 50% O2 - 50% air and 8% desflurane medium flow anesthesia was started with 2 lt/min 50% O2 - 50% air with MAC 1 concentration desflurane.
  Interventions: Other: Medium flow anesthesia
- Minimal flow anesthesia (Experimental): After reaching the MAC 1 value with 4 lt/min 50% O2 - 50% air and 8% desflurane minimal flow anesthesia was started with 0.50 lt/min 50% O2 - 50% air with MAC 1 concentration of desflurane.
  Interventions: Other: Minimal flow anesthesia

INTERVENTIONS:
Other: Medium flow anesthesia — Group MeFA; after reaching the MAC 1 value with 4lt/min 50% O2 - 50% air and 8% desflurane with remifentanil infusion, medium flow anesthesia was started with 2 lt/min 50% O2 - 50% air with MAC 1 concentration desflurane. The vaporizer was closed at the end of the last suture, and the flow was increased to 80% oxygen at 6 lt/min.
  Arms: Medium flow anesthesia
Other: Minimal flow anesthesia — Group MiFA; after reaching the MAC 1 value with 4 lt/min 50% O2 - 50% air and 8% desflurane with remifentanil infusion, minimal flow anesthesia was started with 0.50 lt/min 50% O2 - 50% air with MAC 1 concentration of desflurane. The vaporizer was closed at the end of the last suture, and the flow was increased to 80% oxygen at 6 lt/min.
  Arms: Minimal flow anesthesia

SUMMARY:
The patients were randomized into two groups medium flow anesthesia (MeFA) and minimal flow anesthesia (MiFA). While MeFA received medium flow anesthesia with 2 lt/min, MiFA received minimal flow anesthesia with 0.5 lt/min fresh gas flow. In both groups dynamic compliance values, peak inspiratory pressure (PIP) values, total inhalation anesthetic drug consumption, total remifentanil drug consumption, duration of anesthesia, and duration of surgery were recorded. The FVC, FEV1, and FEV1/FVC values of the patients in both groups were evaluated and noted 24 hours before the operation, after the operation 2nd, 8th, and 24th hours.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* 18-65 years of age, who will undergo elective laparoscopic cholecystectomy surgery

Exclusion Criteria:

* ASA III-IV
* Smokers
* Body mass index (BMI) > 40 kg / m2,
* Patients with cardiovascular system disease
* Chronic respiratory diseases,
* Patients whose pulmonary function tests cannot be applied and who have problems with pulmonary function tests during the examination of the chest disease consultant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Dynamic Compliance assessment | 5th minutes after endotracheal intubation
  Dynamic Compliance will be assessed 5th minutes after endotracheal intubation
Dynamic Compliance assessment | 5th minutes after surgical incision
  Dynamic Compliance will be assessed 5th minutes after the surgical incision
Dynamic Compliance assessment | 10th minutes after surgical incision
  Dynamic Compliance will be assessed 10th minutes after the surgical incision
Dynamic Compliance assessment | 30th minutes after surgical incision
  Dynamic Compliance will be assessed 30th minutes after the surgical incision
Dynamic Compliance assessment | 60th minutes after surgical incision
  Dynamic Compliance will be assessed 60th minutes after the surgical incision
Dynamic Compliance assessment | immediately after the end of the surgical suturing
  Dynamic Compliance will be assessed immediately after the end of the surgical suturing
Peak inspiratory pressure assessment | 5th minutes after endotracheal intubation
  Peak inspiratory pressure will be assessed 5th minutes after endotracheal intubation
Peak inspiratory pressure assessment | 5th minutes after the surgical incision
  Peak inspiratory pressure will be assessed 5th minutes after the surgical incision
Peak inspiratory pressure assessment | 10th minutes after the surgical incision
  Peak inspiratory pressure will be assessed 10th minutes after the surgical incision
Peak inspiratory pressure assessment | 30th minutes after the surgical incision
  Peak inspiratory pressure will be assessed 30th minutes after the surgical incision
Peak inspiratory pressure assessment | 60th minutes after the surgical incision
  Peak inspiratory pressure will be assessed 60th minutes after the surgical incision
Peak inspiratory pressure assessment | immediately after the end of the surgical suturing
  Peak inspiratory pressure will be assessed immediately after the end of the surgical suturing

SECONDARY OUTCOMES:
FEV1 measures assessment | 24 hours before the operation
  FEV1 measures assessment will be assessed 24 hours before the operation
FEV1 measures assessment | 2nd hour after the operation
  FEV1 measures assessment will be assessed 2nd hours after the operation
FEV1 measures assessmentt | 8th hour after the operation
  FEV1 measures assessment will be assessed 8th hours after the operation
FEV1 measures assessment | 24th hour after the operation
  FEV1 measures assessment will be assessed 24th hours after the operation
FVC measures assessment | 24 hours before the operation
  FVC measures assessment will be assessed 24 hours before the operation
FVC measures assessment | 2nd hour after the operation
  FVC measures assessment will be assessed 2nd hour after the operation
FVC measures assessment | 8th hour after the operation
  FVC measures assessment will be assessed 8th hour after the operation
FVC measures assessment | 24th hour after the operation
  FVC measures assessment will be assessed 24th hours after the operation
FEV1/FVC measures assessment | 24 hours before the operation
  FEV1/FVC measures assessment will be assessed 24 hours before the operation
FEV1/FVC measures assessment | 2nd hour after the operation
  FEV1/FVC measures assessment will be assessed 2nd hour after the operation
FEV1/FVC measures assessment | 8th hour after the operation
  FEV1/FVC measures assessment will be assessed 8th hour after the operation
FEV1/FVC measures assessment | 24th hour after the operation
  FEV1/FVC measures assessment will be assessed 24th hour after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Erkan Cem ÇELİK, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Derived] Celik EC, Yayik AM, Aydin ME, Koksal ENM, Disci E, Kerget B, Doymus O, Ahiskalioglu EO, Ahiskalioglu A. Evaluation of lung dynamics and respiratory functions in patients undergoing minimal flow anesthesia: a prospective, randomized controlled trial. Med Gas Res. 2026 Jun 1;16(2):110-115. doi: 10.4103/mgr.MEDGASRES-D-25-00037. Epub 2025 Aug 18. PMID 40826933